CLINICAL TRIAL: NCT06581445
Title: Psychophysiological Effects of Birdsongs on Sadness: Compared With Music Between Depressed and Non-Depressed Participants
Brief Title: Psychophysiological Effects of Birdsongs VS Music
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Shulin Chen, Professor, Zhejiang University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Effects of Birdsongs
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Sadness
Keywords: Birdsongs; music; sadness; depressive symptoms; psychophysiological effects
MeSH Terms: conditions — Depression | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were told that this experiment was to examine the different effects between video stimuli and audio stimuli.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depressed group (Experimental): The participants were categorized into two groups using the Patient Health Questionnaire (PHQ-9) and the 17-item Hamilton Depression Rating Scale (HAM-D). PHQ-9 is a self-report scale. PHQ-9 scores of 5 or higher represent mild and severe depression, while PHQ-9 scores of lower than 5 mean normal condition. HAM-D is a scale administered by a healthcare professional. The cut-off point of the HAM-D scale is 8, which divides normal conditions from depressive conditions. The participants first completed PHQ-9. For those with PHQ-9 scores of 5 or higher, the trained researchers interviewed them and rated their severity of depression on the HAM-D. The participants first completed PHQ-9.
  For those with PHQ-9 scores ≥ 5, the trained researchers interviewed them and rated their severity of depression on the HAM-D. Those with HAM-D scores > 8 were classified into the depressed group.
  Interventions: Behavioral: Birdsongs; Behavioral: Music
- Non-depressed group (Experimental): Those with PHQ-9 scores < 5 or HAM-D scores ≤ 8 were classified into the non-depressed group.
  Interventions: Behavioral: Birdsongs; Behavioral: Music

INTERVENTIONS:
Behavioral: Birdsongs — The participants listened to a clip of birdsongs from laughing thrushes.
Behavioral: Music — The participants listened to a cheerful Cuckoo Waltz music.

SUMMARY:
The main goal of this study is to learn the psychophysiological effects of birdsongs on sadness. The main questions it aims to answer are:

1. Can birdsongs alleviate sadness in a short term?
2. Can birdsongs have greater impact on sadness than music?
3. Can birdsongs alleviate sadness for both non-depressed and depressed participants?

Researchers will compare birdsongs to music (a active control) to see if birdsongs works to reduce sadness and also examined the psychophysiological effects of birdsongs in depressed and non-depressed participants.

Participants will:

go through the following stages: baseline, neutral control, 1st sadness induction, 1st intervention, calculation task, 2nd sadness induction, and 2nd intervention.

DETAILED DESCRIPTION:
During the baseline phase, participants were instructed to sit quietly and relax. For the neutral control, they viewed an informative video demonstrating the process of plastic injection molding. As for the sadness induction, they were presented with sad film clips from either Hachi: A Dog's Tale or My Brother and Sister. The order of the sad videos was randomized across participants. The intervention stages involved listening to either the cheerful Cuckoo Waltz music or a clip of birdsongs from laughing thrushes. The order of the interventions was randomized as well. The calculation task was employed as a distracter, enabling participants to return to a neutral state. Except for the computational task, the remaining six phases each had a duration of 6 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years
* Right-handed
* No recent illness or medication use
* No history of neurological or psychiatric disorders
* Normal or corrected-to-normal visual acuity (myopic participants wore glasses)
* Normal hearing

Exclusion Criteria:

* Incapable of giving written informed consent to this study
* Acute high suicide risk at baseline assessment
* Psychosis

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Self-Assessment Manikin (SAM) | Immediately after the baseline, immediately after the neutral control, immediately after each sadness induction, and immediately after each intervention.
  The SAM scale is a brief and widely used tool for assessing emotional states. The scale is a nonverbal self-report measure of emotion, using a set of cartoon-like manikins. The manikins illustrate nine intensity levels for valence (1 = unpleasant; 9 = pleasant), arousal (1 = calm, 9 = excited), and dominance (1 = controlled; 9 = controlling).
Revision of Positive Affect and Negative Affect Scale (PANAS-R) | Immediately after the baseline, immediately after the neutral control, immediately after each sadness induction, and immediately after each intervention.
  The PANAS is another widely used scale to measure mood or emotion. The Chinese version of PANAS is comprised of 18 items, with 9 items measuring positive affect (e.g., joyful, inspired) and 9 items measuring negative affect (e.g., sad, fearful). Because participants were required to report their feelings repeatedly in this study, 18 items would be too long and tiresome. The 18 items plus "calmness" were used as 19 options for participants to choose. They needed to select one of the emotion words to tag their strongest emotion for the stage that they had just experienced. This revision of PANAS allowed us to capture the specific emotion type.
Mean of Normal-to-Normal Intervals (MeanNN) | Throughout the whole experiment, an average of 6 minutes for each stage.
  MeanNN refers to the average duration between consecutive normal heartbeats, also named inter-beat interval. A higher MeanNN indicates a lower heart rate.
Standard Deviation of Normal-to-Normal Intervals (SDNN) | Throughout the whole experiment, an average of 6 minutes for each stage.
  SDNN measures the overall variability of heart rate. Higher SDNN values indicate greater variability.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China